CLINICAL TRIAL: NCT03355352
Title: Observational Study of Analgesia and Cost-efficiency of Analgetic Medication Pumps (Zalviso and PCA-syringe Pump) After Urogenital Intervention at the Clinical Daily Routine
Brief Title: Observational Study of Analgesia and Cost-efficiency of Analgetic Medication Pumps (Zalviso and PCA-syringe Pump (PCA=Patient Controlled Analgesia)) After Urogenital Intervention at the Clinical Daily Routine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: 277/2017BO1
Record Dates: First submitted 2017-11-20; First posted 2017-11-28 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Analgesic Quality; Mobility
Keywords: Zalviso; sufentanyl; PCA; Dipidolor
MeSH Terms: interventions — Sufentanil

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients treated with conventional i.v. PCA
- Patients treated with Zalviso
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Sufentanil — Sufentail sublingual 15ug nanopills
  Groups: Patients treated with Zalviso

SUMMARY:
The observational study will check if there is a difference in the postoperative care of patients with urogenital intervention while using the standard PCA-syringe pump or using the Zalviso sufentanyl sublingual analgetic system.

The study will exactly examine, using questionaire for the patient, the medical stuff (nurses and anesthesiologist) the difference in the analgetic quality, the difference of the patients' mobility while being treated with one of the analgetic system and if there is a difference in the cost-efficiency.

We want to examine 50 Patients in each group. The studies should be finished in about one year.

ELIGIBILITY:
Inclusion Criteria:

* Patients after urological interventions with no indication of an periduralanästesia
* Patients compliant for a PCA system, and complied with the analysis of their data

Exclusion Criteria:

* F03 dementia
* F10.2 dependence syndrome alcohol
* F11.2 dependence syndrome opioids
* F12.2 dependence syndrome cannabinoids
* F13.2 dependence syndrome sedatives and hypnotics
* F14.2 dependence syndrome cocaine
* F15.2 dependence syndrome coffin
* F.16.2 dependence syndrome hallucinogens
* F22 schizophrenia
* F41.1 generalized anxiety disorder

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients at the teaching hospital of university tuebingen which get an surgical urological intervention and which correspond with the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-08-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
analgesic quality | 1 year
  Recording of the analgesic quality measured by the request of more analgesic postoperative while being treated with the conventional PCA or the Zalviso system.
mobility | 1 year
  Recording of the patients mobility postoperative while being treated with the conventional PCA or the Zalviso system.

SECONDARY OUTCOMES:
medical cost efficiency | 1 year
  Comparison of the cost efficiency of both systems

CONTACTS AND LOCATIONS:
Locations (1):
- University Tuebingen, clinic of anästhesiology and intensiv care, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No